CLINICAL TRIAL: NCT04996420
Title: Goal Directed Fluid Management vs Liberal Fluid Regimen Based on Mean Arterial Pressure in Patients Undergoing Spinal Anesthesia for Primary Elective Hip Arthroplasty: a Randomized, Prospective, Controlled Study."
Brief Title: Goal Directed Fluid Therapy Versus Liberal Fluid Regimen in Primary Elective Hip Artrhoplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: change in surgical technique (lateral approach vs anterior approach for hip arthroplasty, determining a change in patient intraoperative positioning)
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Emospin 2
Record Dates: First submitted 2020-01-29; First posted 2021-08-09 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2021-07

CONDITIONS: Arthroplasty, Replacement, Hip; Anesthesia, Spinal; Hemodynamic Monitoring; Crystalloid Solutions

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Clearsight (Experimental): hemodynamic monitoring and goal directed fluid therapy guided by clearsight
  Interventions: Device: Clearsight non invasive hemodynamic monitoring
- Control (Other): hemodynamic monitoring blinded and silenced, no goal directed fluid therapy. Fluid therapy based on clinical evaluation and mean arterial pressure by non-invasive monitoring
  Interventions: Device: Clearsight non invasive hemodynamic monitoring

INTERVENTIONS:
Device: Clearsight non invasive hemodynamic monitoring — Goal directed fluid therapy fuided by Clearsight monitoring

SUMMARY:
Patients undergoing elective primary total hip replacement and spinal anesthesia may encounter significant hemodynamic instability.

The study is a randomized controlled type and is aimed at comparing how perioperatory hypotension and fluid regimen are managed using Clearsight non invasive monitoring system or PAM monitoring.

The primary endpoint is to evaluate total duration of hypotension, defined as a MAP < 65 mmHg, calculated during all the perioperatory time.

Fifty-eight patients, aged 50-80 years, with an American Society of Anaesthesiologists' (ASA) score I, II and III were enrolled and split in two groups (Clearsight and control group). Patients were monitored both with the EV1000 platform, the Clearsight finger-cuff and MAP monitoring. Depending on the group, the fluid regimen was a goal directed fluid therapy or a liberal fluid regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-80 years
* ASA I, II or III
* primary elective hip arthroplasty

Exclusion Criteria:

* spinal anesthesia contraindications
* periferical vasculopaty
* other diseases which indicates better an invasive monitoring by radial artery cannulation
* atrial fibrillation
* denial or inability to provide informed consent

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2020-11-22 (Actual); Study Completion 2020-11-22 (Actual)

PRIMARY OUTCOMES:
total perioperative hypotension time defined by a mean arterial pressure < 65mmHg, from arrival in the anesthesia induction room to resolution of spinal block in Recovery Room (i.e. up to 8 hours) | from arrival in the anesthesia induction room to resolution of spinal block in Recovery Room

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Bonarelli, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- IORizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided